CLINICAL TRIAL: NCT05761041
Title: Effectiveness of Silver Diamine Fluoride Versus Sodium Fluoride Varnish With Parental Behavior Modification for Arresting Early Childhood Caries: A Randomized Clinical Trial
Brief Title: Silver Diamine Fluoride Versus Sodium Fluoride Varnish With Parental Behavior Modification in Arresting Early Childhood Caries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Science, Technology & Innovation Funding Authority (STDF) (Unknown)
Responsible Party: Principal Investigator, randa hassan abdelsamea yassin, Teaching Assistant, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0272 - 07 /2021
Record Dates: First submitted 2023-02-14; First posted 2023-03-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Early Childhood Caries
Keywords: ECC; 38% SDF; 5% NaF; Motivational Interviewing; Preschoolers
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naf + MI (Experimental): Sodium Fluoride Varnish 5% (Applied biannually) + two MI sessions: baseline face-to-face session and phone call after 3months.
  Interventions: Drug: Sodium Fluoride Varnish (5%); Behavioral: Motivational Interviewing
- SDF (Active Comparator): Silver Diamine fluoride 38% (Applied biannually)
  Interventions: Drug: SDF

INTERVENTIONS:
Drug: Sodium Fluoride Varnish (5%) — Applied at baseline
  Arms: Naf + MI
Behavioral: Motivational Interviewing — Two MI sessions: face-to-face at baseline and phone call at 3 months
  Arms: Naf + MI
Drug: SDF — Applied bianually
  Arms: SDF

SUMMARY:
Arresting dental caries using silver diamine fluoride (SDF) has gained attention recently for the management of early childhood caries (ECC). However, black staining is one of its drawbacks. A possible affordable alternative can be Sodium Fluoride (NaF) supported with good oral hygiene induced by parental Motivational Interviewing (MI).

The trial aims to compare the impact of SDF versus NaF supported by MI on lesion activity in preschool children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged ≤ 4 years old.
2. The presence of at least one active carious lesion on a primary tooth, with scores 3 and higher (according to the International Detection and Assessment System- ICDAS II)
3. Children whose caregivers have means of communication (mobile phones).
4. Completion of an informed consent to participate in the study.

Exclusion Criteria:

1. Children reporting spontaneous or elicited pain from caries or showing any signs of pulpal infection, swelling and/or abscess.
2. Parental refusal to participate in the study.
3. Allergy or sensitivity to silver or any of the materials included in the study.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Caries Arrest | 6 months
  Percentage of arrested carious lesions

SECONDARY OUTCOMES:
Caries Increment | 6 months
  Number of new carious lesions will be assessed using decayed, missing (due to caries), and filled primary tooth surface index (dmfs)
Parental satisfaction | Baseline and 6 months
  Parents will be asked if application was an easy process, pain free for their child and taste is acceptable. Answers will be on a 5 point Likert scale (Strongly agree, Agree, Neutral , Disagree, Strongly disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yassin R, Amer H, Tantawi ME. Effectiveness of silver diamine fluoride versus sodium fluoride varnish combined with mother's motivational interviewing for arresting early childhood caries: a randomized clinical trial. BMC Oral Health. 2023 Oct 4;23(1):710. doi: 10.1186/s12903-023-03456-3. PMID 37789300